CLINICAL TRIAL: NCT02965157
Title: Pilot Study of Anti-CD20-CAR-engineered T Cells in Patients With Chemotherapy Resistant or Refractory CD20+ Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Biohealthcare Biotechnology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EY201605-19
Record Dates: First submitted 2016-08-31; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CART20 (Experimental)
  Interventions: Biological: CART20

INTERVENTIONS:
Biological: CART20

SUMMARY:
Chimeric antigen receptor (CAR) T cells targeting CD20 will be evaluated for safety and efficacy in patients with CD20+ B cell lymphoma. The CAR consists of a CD20 targeting antibody scFv with two intracellular signaling domains derived from CD3 zeta and CD28. Autologous T cells will be gene-engineered with the CAR gene using a retrovirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory CD20+ B-cell lymphoma.
2. Measurable disease.
3. Performance status ECOG 0-2.
4. Age:18-65.
5. Fertile females/males must consent to use contraceptives during participation of the trial.
6. Signed informed consent

Exclusion Criteria:

1. Any significant medical or psychiatric illness that would prevent the patient from giving informed consent or from following the study procedures.
2. Patients with primary CNS lymphoma.
3. Known human immunodeficiency virus (HIV) infection.
4. Active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection).
5. Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient.
6. Treatment with an investigational product within 30 days prior to enrollment, or at least 5 half lives of that drug, which is longest.
7. Patients that do not consent to that tissue and blood samples are stored in a biobank.
8. Pregnancy.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences Tumor Hospital, Beijing, China